A Multi-center Clinical Study on the Efficacy and Safety of Kuntai

Capsule Alone and in Combination With Hormones in the Treatment

of Early-onset Hypoovarian Function

NCT05021094

**Date: August 4, 2021** 

Statistical analysis

The case observation form completed by the test center was reviewed and returned by

the project team of Shanghai Haitian Pharmaceutical Technology Development Co.,

Ltd., and the data was processed by a statistical analyst. The data in the case report

form is entered in two copies, and the database is locked after verification and

confirmation. SPSS26.0 software was used for statistical analysis. The full analysis

set (FAS) and the per-protocol set (PPS) were used for effectiveness analysis, and the

safety data set (SS) was used for safety analysis. Measurement data were expressed as

mean  $\pm$  standard deviation (x  $\pm$  s), multiple time points were compared by repeated

measures analysis of variance, and pairwise comparisons were by Bonferroni test;

enumeration data were expressed by the number of cases or percentages, and  $\chi^2$  was

used.Test for statistical comparison.P<0.05 indicated that the difference was

statistically significant.